CLINICAL TRIAL: NCT07218445
Title: The Effect of Tirzepatide on Menopausal Vasomotor Symptoms and Biological Aging in Post-menopausal Women With Obesity: A Pilot Study
Brief Title: The Effect of Tirzepatide on Menopausal Vasomotor Symptoms and Biological Aging in Post-menopausal Women With Obesity
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Chrisandra L. Shufelt, MD, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 25-001692
Record Dates: First submitted 2025-10-03; First posted 2025-10-20 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Obesity; Menopause Hot Flashes
Keywords: Hot flashes; menopause; Tirzepatide; GLP
MeSH Terms: conditions — Obesity; Hot Flashes | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tirzepatide (Experimental): Participants will receive tirzepatide for 24 weeks, in addition to standard lifestyle modification recommendations
  Interventions: Drug: Tirzepatide
- Placebo (Placebo Comparator): Participants will receive a placebo for 24 weeks, in addition to standard lifestyle modification recommendations
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirzepatide — Tirzepatide will be administered with a starting dose of 2.5 mg weekly, subcutaneously injected. The dose will increase by 2.5 mg every 4 weeks until reaching 15 mg.
  Participants will be asked to follow lifestyle interventions:
  * Low-calorie diet based on their predicted by Harris Benedict resting energy expenditure minus 500 kcal per day
  * Physical activity: a goal of 10,000 steps or more per day
  * Exercise: a goal of 150 minutes or more of moderate-intensity aerobic activity (cardiovascular exercise) per week
  * Limited consumption of liquid calories (i.e. sodas, juices, alcohol, etc.).
  Arms: Tirzepatide
Drug: Placebo — A placebo for Tirzepatide will be administered with a starting dose of 2.5 mg weekly, subcutaneously injected. The dose will increase by 2.5 mg every 4 weeks until reaching 15 mg.
  Participants will be asked to follow lifestyle interventions:
  * Low-calorie diet based on their predicted by Harris Benedict resting energy expenditure minus 500 kcal per day
  * Physical activity: a goal of 10,000 steps or more per day
  * Exercise: a goal of 150 minutes or more of moderate-intensity aerobic activity (cardiovascular exercise) per week
  * Limited consumption of liquid calories (i.e. sodas, juices, alcohol, etc.).
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effect of tirzepatide on vasomotor symptoms and on measures of biological aging.

ELIGIBILITY:
Inclusion Criteria

* Postmenopausal women defined as 12 months of spontaneous amenorrhea, or 6 months of spontaneous amenorrhea with serum follicle-stimulating hormone (FSH) levels > 40 mIU/ml, or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy.
* Age 46-60 years old.
* BMI ≥30 kg/m2 or BMI ≥27 kg/m2 in the presence of adiposity-associated diseases (hypertension, dyslipidemia, obstructive sleep apnea, cardiovascular disease).
* Presence of bothersome hot flashes (≥ 28 episodes per week and of sufficient severity to prompt patients to seek therapeutic interventions).
* Hot flashes must be present for >30 days prior to study entry.
* Ability to participate in all portions of the study, including willingness to self-inject drug
* Provided informed consent to be part of the study.
* Willingness and capability to follow a hypocaloric diet, consisting of an energy deficit of approximately 500 kcal/day compared to baseline total energy expenditure, and composed of 30% from fat, 20% from protein, and 50% of carbohydrate. In addition to performing at least 150 min/week of physical activity

Exclusion Criteria

* Current treatment with menopausal hormone therapy.
* Any current (past 4 weeks) or planned use of:

  * Estrogen-containing contraceptive methods or menopausal hormone therapy (oral, transdermal, high dose vaginal ring, injection, pellets).
  * Vaginal estrogen.
  * Androgens.
  * Progestogens.
* Current treatment for menopausal symptoms with cognitive behavioral therapy and/or hypnosis.
* Current use of fezolinetant.
* Menopause as a result of cancer treatments.
* Impaired renal function (GFR ≤30 ml/min/1.73 m²).
* Thyroid-stimulating hormone ≥7 with low free T4.
* 10-year ASCVD risk > 7.5%.
* Active inflammatory, autoimmune, infectious, hepatic, gastrointestinal, malignancy, or uncontrolled psychiatric disease.
* >5% change in weight during the 3 months prior to screening and, or eight fluctuation of ≥20 pounds within the past 6 months (self-report).
* Other obesity medication used within the past 3 months.
* History of bariatric surgery. Prior or planned surgical treatment for obesity (excluding liposuction or abdominoplasty performed > 1 year before screening).
* Past or intended endoscopic and/or device-based therapy or removal within last six months.
* Current or recent (within 3 months) use of medications that may cause weight gain, including tricyclic antidepressants, atypical antipsychotics, and mood stabilizers.
* Current or recent (within 3 months) use of chronic systemic glucocorticoid therapy for over 2 weeks within the past 3 months.
* Contraindications to GLP-1 receptor agonist therapy as per Tirzepatide (Zepbound ®) label, including a personal or family history of medullary thyroid carcinoma; a history or diagnosis of multiple endocrine neoplasia syndrome type 2; known hypersensitivity to tirzepatide or any of its excipients.
* Currently enrolled in another clinical study involving an investigational product, or participated in one and received treatment (active or placebo) in the last 30 days.
* Planned surgical procedures requiring general anesthesia or sedation during the study or within 2 weeks following the last dose of study drug.

Ages: 46 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2027-09-18 (Estimated); Study Completion 2027-09-18 (Estimated)

PRIMARY OUTCOMES:
Change in Vasomotor Symptoms Frequency | Baseline, 24 weeks
  Change in the frequency of self-reported daily average vasomotor symptoms from baseline to 24 weeks. Vasomotor symptoms will be captured for 2 weeks at baseline and 2 weeks at the end of the study.
Change in Vasomotor Symptom Severity | Baseline, 24 weeks
  Change in self-reported daily vasomotor symptom severity from baseline to 24 weeks. Vasomotor symptoms will be captured for 2 weeks at baseline and at the end of the study. Severity will be classified as follows:
  Mild, sensation of heat without sweating/dampness; Moderate: sensation of heat with sweating/dampness, but able to continue current activity. May briefly fan yourself; Severe: sensation of intense heat with sweating causing disruption of current activity.
Aging Biomarkers: Cellular Senescence Markers in Plasma | 24 weeks
  Cellular senescence markers are measured in plasma samples to assess biological aging and cellular stress. These markers may include proteins associated with the senescence-associated secretory phenotype (SASP). Quantification is performed using immunoassays. Higher levels of senescence markers indicate increased cellular senescence.
Difference between biological and chronological age | 24 weeks
  Epigenetic clocks estimate biological age by analyzing DNA methylation patterns at specific CpG sites across the genome. Biological age estimates are compared to chronological age to assess aging acceleration or deceleration. Biological age greater than chronological age indicates accelerated biological aging and potential increased risk of morbidity and mortality. Primary measure is the difference (ΔAge) between biological and chronological ages = reported in years.

SECONDARY OUTCOMES:
Change in Reactive hyperemic index | Baseline, 12 weeks and 24 weeks
  Vascular function will be measured using the EndoPAT device to assesses reactive hyperemia index (RHI) from baseline to week 24 on treatment or placebo. RHI is automatically calculated through a computer algorithm by following the equation: [(tested arm-post occlusion/tested arm-baseline)/(control arm-post occlusion/control arm-baseline)] × baseline correction factor. Endothelial dysfunction is defined as having an RHI ratio of equal or less than 1.67.
Change in Augmentation Index percentage | Baseline, 12 weeks, and 24 weeks
  Augmentation Index (AIx): AIX uses applanation tonometry of the radial artery pulse, calibrated to resting brachial systolic and diastolic pressures (SphygmoCor XCEL, Medtronic, Minneapolis, MN). Aortic systolic, diastolic, and pulse pressures will be derived from a synthesized aortic waveform using a validated mathematical transfer function. Augmentation pressure, reflecting the difference between aortic systolic pressure and the inflection point caused by the reflected wave, is influenced by arterial stiffness as well as factors like heart rate and ejection dynamics. AIx is calculated as augmentation pressure divided by aortic pulse pressure × 100%, adjusted to a heart rate of 75 bpm (AIx@75 bpm). Measurements will be performed in duplicate and averaged.
Change in Pulse Wave Velocity | Baseline, 12 weeks, and 24 weeks
  SphygmoCor estimates central arterial stiffness by calculating the speed at which the pressure wave travels between the carotid and femoral arteries using applanation tonometry and reported as the pulse wave velocity (PWV); PWV m/s
Change in Cardiometabolic Parameters: Blood Pressure | Baseline, 24 weeks
  Change in cardiometabolic parameters including blood pressure from baseline to week 24 on treatment or placebo. Measured in mmhg
Change in Cardiometabolic Parameters: Fasting Glucose | Baseline, 24 weeks
  Change in cardiometabolic parameters including fasting glucose from baseline to week 24 on treatment or placebo. Measured in mg/dL
Changes in Cardiometabolic Parameters: HbA1C | Baseline, 24 weeks
  Change in cardiometabolic parameters including HbA1C from baseline to week 24 on treatment or placebo. Measured in %
Changes in Cardiometabolic Parameters: Lipoprotein profile | Baseline, 24 weeks
  Change in cardiometabolic parameters including Lipoprotein profile from baseline to week 24 on treatment or placebo. Measured in mg/dL
Changes in Cardiometabolic Parameters: hsCRP | Baseline, 24 weeks
  Change in cardiometabolic parameters including hsCRP from baseline to week 24 on treatment or placebo. Measured in mg/L
Change in Physical Function Measure: Short Physical Performance Battery (SPPB) score. | Baseline, 24 weeks
  The SPPB is a standardized test that evaluates lower extremity function using three components: balance tests (standing in various positions), gait speed (walking a short distance), and chair stand (repeated standing from a seated position). Each component is scored from 0 to 4; the total score ranges from 0 to 12. Higher scores represent better physical function
Change in Physical Function Measure: Modified Clinical Test of Sensory Interaction in Balance (mCTSIB) performed on the Rehabilitation Artificial Physical Intelligence Database (RAPID) foot pressure mat | Baseline, 24 weeks
  The mCTSIB assesses balance under four sensory conditions: eyes open/closed on firm and foam surfaces. Testing is performed while standing on the RAPID foot pressure mat, which captures center of pressure and postural sway data. The primary measure is average sway area of the four sensory conditions. The sway area is the area which is required to correct equilibrium, representing the total area covered by postural sway, measured in square centimeters (cm²).
Change in Physical Function Measure: Standing Chest Throw Test with a 2-kg Weighted Ball using Motion Sensor Technology (MST) | Baseline, 24 weeks
  This test evaluates upper body muscular power. Participants perform a two-handed chest throw of a 2-kg medicine ball from a standing position. The MST is used to record throw distance, velocity, and related performance metrics. The primary measure is Peak Power Score (W).
Change in Physical Function Measure: Chair-to-Stand Tests using Motion Sensor Technology (MST) | Baseline, 24 weeks
  This test assesses lower body strength and function. Participants are instructed to stand up from a chair and sit back down five times without using their arms. The MST measures movement dynamics. The primary measure is peak power score (W).
Change in Physical Function Measure: Six-Minute Walk Test (6MWT) | Baseline, 24 weeks
  The 6MWT is a standardized submaximal exercise test used to assess functional aerobic capacity. Participants are instructed to walk as far as possible in six minutes along a flat, straight course. The total distance walked is recorded in feet. Longer walking distances indicate better aerobic capacity and endurance.
Change in Physical Function Measure: Hand Grip Strength using a Hydraulic Hand Dynamometer | Baseline, 24 weeks
  Participants are instructed to squeeze the dynamometer with maximum effort, measured in kilograms. The highest value from multiple trials is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Chrisandra Shufelt, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials/cls-20589486